CLINICAL TRIAL: NCT03037112
Title: Resetting the Default: Improving Provider-patient Communication to Reduce Antibiotic Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Heartland Primary Care of Sunflower Medical Group (Unknown); Washington University School of Medicine (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kathy Goggin, Ernest L. Glasscock, MD, Chair in Pediatric Education and Research, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PCORI150731759
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Communication; Anti-Bacterial Agents; Decision Making; Personal Satisfaction
MeSH Terms: conditions — Communication; Personal Satisfaction | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Providers will be randomly assigned to the education or communication skills intervention study arms. Both groups will receive identical training on the appropriate prescribing of antibiotics for ARTIs, but only those in the communication intervention will receive additional training on communication skills. Once providers have been randomized and trained, eligible patients will be enrolled and exposed to one of the interventions based on the provider they see for their visit. Patients will not be informed of their provider's study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Active Comparator): All providers will receive identical training on the appropriate prescribing of antibiotics for ARTIs in a 20 minute presentation. Follow up refresher video clips will also be available for all providers to view at their convenience throughout the study. Parents in both arms will receive identical high quality education on the pros and cons of antibiotics and tips for communicating with their provider.
  Interventions: Behavioral: Education
- Communication Skills (Active Comparator): Providers randomized to the communication intervention will receive additional training on communication skills in a 40 minute communication skills training session. This training session will include good and bad communication examples, training on positive and negative behavioral framing, and education regarding key drivers of patient satisfaction.
  Interventions: Behavioral: Communication Skills

INTERVENTIONS:
Behavioral: Education — The first intervention is an educational intervention regarding appropriate diagnosis and treatment of common respiratory infections. This education will be delivered in an interactive lecture format for providers with follow up short informational video clips available over the course of the project.
  Arms: Education
Behavioral: Communication Skills — The second intervention is an education plus communication skills training intervention. This training session will include identical antibiotic education training, good and bad communication examples, training on negative behavioral framing, and education regarding key drivers of patient satisfaction. Additionally providers will be informed of parent's desire for antibiotics rating prior to their consultation with the patient.
  Arms: Communication Skills

SUMMARY:
Antibiotic overuse and misuse contributes to the development of antibiotic resistant infections and adverse drug reactions. The majority of all antibiotic prescribing occurs in outpatient settings; most of which are for respiratory illnesses. It is estimated that 50% of these prescriptions are unnecessary. The most important factor that leads to overprescribing is inadequate parent-provider communication. This study will recruit providers and eligible parents of children 1-5 years of age. Parents in both arms will receive identical brief antibiotic education via tablet computers. Providers will be randomized to the parent-provider education or communication skills intervention arm and trained accordingly. Parent data will be collected via a tablet computer RedCap survey administered in the exam room prior and immediately following the child's visit. Additional data will be garnered from the medical record (antibiotic prescribing) and a 2-week follow-up telephone call with parents (re-visits and adverse drug reactions).

DETAILED DESCRIPTION:
Significance: Antibiotic overuse and misuse contribute to the development of antibiotic resistant infections that kill at least 23,000 Americans and cause an additional 2 million infections annually. If left unchecked, antibiotic resistant infections are estimated to cause 10 million deaths worldwide by 2050. Antibiotic associated adverse drug reactions (e.g., rash, diarrhea, nausea, and vomiting) also result in over 140,000 Emergency Department visits annually.

The majority of all antibiotic prescribing occurs in outpatient settings where children receive 49 million prescriptions annually. Over 70% of these are for respiratory infections and nearly 8.5 million of these prescriptions are inappropriate (i.e., either an unnecessary broad-spectrum antibiotic or to treat a viral illness). There are many factors that lead to overprescribing, but chief among them is inadequate parent-provider communication.

Innovation: This study is the first US multi-site randomized controlled trial comparing the effectiveness an education vs. communication skills provider intervention to stimulate high quality parent-provider communication and judicious use of antibiotics.

Approach: 1,600 eligible parents (or caregivers) of children between the ages of 1 and 5 will be enrolled and exposed to one of the interventions based on the provider they see for their visit. English and Spanish speaking parents will be recruited from the Children's Mercy Hospital Primary Care Clinic (CMH PCC) in Kansas City, Missouri and the Heartland Primary Care Clinics in Kansas City, KS and Lenexa, KS. Parents in both arms will receive identical brief negatively behavioral framed antibiotic education via tablet computers. Providers will be randomized to the parent-provider education or communication skills intervention arm and trained accordingly. The primary outcome is rate of inappropriate antibiotic prescribing. Secondary outcomes are parental ratings of shared decision-making and satisfaction, re-visits and adverse drug reactions. Data will be collected via a tablet computer administered RedCap survey administered in the exam room prior and immediately following the child's visit. Additional data will be garnered from the medical record (antibiotic prescribing) and a 2-week follow-up telephone call with parents (re-visits and adverse drug reactions).

Public Health Impact: This study could have significant public health implications and meet the goals outlined in the 2014 Executive Order on Combating Antibiotic Resistance, which seeks to slow the emergence of resistant bacteria and prevent the spread of resistant infections through the judicious and appropriate use of antibiotics.

ELIGIBILITY:
Inclusion Criteria: \

* Parent or guardian of a child 1-5 years of age with suspected respiratory tract infection who are English or Spanish speaking

Exclusion Criteria:

* Parents of children who require hospitalization
* Received antibiotics in the last 30 days
* Have concurrent bacterial infection, an immune compromising condition or chronic medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Inappropriate antibiotic use | 18 months
  Patient medical records will be reviewed 2 weeks after the visit to determine the clinical diagnosis and whether or not antibiotics were given. Determination will be made regarding the appropriateness of the diagnosis and prescribing using current clinical practice guidelines.

SECONDARY OUTCOMES:
Revisits | 18 months
  All parents will be called 2 weeks following the initial visit to determine if any revisits to the same office or to another health care facility were made after the initial visit for either clinical worsening or lack of clinical improvement, or due to an adverse drug reaction.
Adverse drug reactions | 18 months
  All parents will be called 2 weeks following the visit to determine if the patient developed an adverse drug reaction to antibiotics.
Shared decision-making | 18 months
  Parents will rate the quality of the shared decision-making using validated survey instruments
Parent Satisfaction with visit | 18 months
  Parents will rate the their satisfaction with the visit using validated measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Goggin, PhD, Principal Investigator — Childrens Mercy Hospital; Jason G. Newland, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Heartland Primary Care, Kansas City, Kansas
  - Heartland Primary Care, Lenexa, Kansas
  - Children's Mercy Pediatric Care Clinic, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Yes
We will create a clean, de-identified copy of our final dataset that will be available to other researcher groups, upon request, within 9 months of the end of the final year of funding. Prior to data sharing, we will remove or convert all identifying information (date of birth will be converted to age and other identifiers will be removed). There may remain the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users under a data-sharing agreement.

REFERENCES:
- [Derived] Goggin K, Hurley EA, Lee BR, Bradley-Ewing A, Bickford C, Pina K, Donis de Miranda E, Yu D, Weltmer K, Linnemayr S, Butler CC, Newland JG, Myers AL. Let's Talk About Antibiotics: a randomised trial of two interventions to reduce antibiotic misuse. BMJ Open. 2022 Nov 21;12(11):e049258. doi: 10.1136/bmjopen-2021-049258. PMID 36410835
- [Derived] Goggin K, Hurley EA, Bradley-Ewing A, Bickford C, Lee BR, Pina K, De Miranda ED, Mackenzie A, Yu D, Weltmer K, Linnemayr S, Butler CC, Miller M, Newland JG, Myers AL. Reductions in Parent Interest in Receiving Antibiotics following a 90-Second Video Intervention in Outpatient Pediatric Clinics. J Pediatr. 2020 Oct;225:138-145.e1. doi: 10.1016/j.jpeds.2020.06.027. Epub 2020 Jun 15. PMID 32553835
- [Derived] Goggin K, Bradley-Ewing A, Myers AL, Lee BR, Hurley EA, Delay KB, Schlachter S, Ramphal A, Pina K, Yu D, Weltmer K, Linnemayr S, Butler CC, Newland JG. Protocol for a randomised trial of higher versus lower intensity patient-provider communication interventions to reduce antibiotic misuse in two paediatric ambulatory clinics in the USA. BMJ Open. 2018 May 9;8(5):e020981. doi: 10.1136/bmjopen-2017-020981. PMID 29743330